CLINICAL TRIAL: NCT07298707
Title: A Multicenter Study on Cervical Cytology DNA Methylation for Screening and Follow-up of Endometrial Lesions
Brief Title: Cervical Cytology DNA Methylation for Endometrial Lesion Screening and Follow-up
Acronym: EndoMethy-V
Status: Not yet recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Beijing Tiantan Hospital (Other); The Third Xiangya Hospital of Central South University (Other); Beijing Chuiyangliu Hospital (Other Government); Beijing Sixth Hospital (Unknown)
Responsible Party: Principal Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Other Study IDs: K9518; ZS-2740 (Other Grant/Funding Number: Beijing Natural Science Foundation)
Record Dates: First submitted 2025-12-09; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Endometrial Neoplasms; DNA Methylation; Cervical Smears; Early Detection of Cancer; Endometrial Hyperplasia
MeSH Terms: conditions — Endometrial Neoplasms; Endometrial Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endometrial Cancer Risk Cohort: This is a prospective, observational cohort of women at medium-to-high risk for endometrial cancer. All participants undergo baseline cervical cytology sampling for DNA methylation testing (CISENDO) and diagnostic hysteroscopy. Follow-up strategy is stratified based on initial methylation results and risk factors, with some receiving repeat methylation testing and/or hysteroscopy at 6 and 12 months, and others receiving methylation testing only.

SUMMARY:
The goal of this observational study is to evaluate the accuracy of a novel molecular test for screening and monitoring endometrial lesions in women at medium-to-high risk for endometrial cancer.

The main questions it aims to answer are:

* What is the sensitivity and specificity of the CISENDO test (a DNA methylation test on cervical cytology samples) for detecting histologically confirmed endometrial intraepithelial neoplasia (EIN) or invasive endometrial cancer?
* How do DNA methylation levels change during the follow-up of endometrial lesions? Researchers will compare the results of the CISENDO test to the results from the standard diagnostic procedure (hysteroscopy with histology) to see if the molecular test can reliably identify high-risk lesions and track disease progression.

Participants will:

* Provide a residual liquid-based cervical cytology sample for the CISENDO test.
* Undergo a standard diagnostic hysteroscopy examination (with or without biopsy) for comparison.
* Some participants will return for follow-up visits at 6 and 12 months for repeat methylation testing and/or hysteroscopy to monitor their condition.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be 18 years of age or older.
2. Participants must possess medium-to-high risk factors for endometrial cancer as defined by Chinese consensus guidelines and are scheduled for hysteroscopic evaluation; OR are currently undergoing conservative treatment (e.g., progesterone therapy or endometrial ablation) for endometrial lesions, and have not received chemotherapy.
3. Participants must be capable and willing to provide written informed consent.
4. Participants must be willing to undergo at least one follow-up assessment within 1 year.
5. Participants must have an intact cervix (a history of LEEP or conization is acceptable).

Exclusion Criteria:

1. Current treatment for any gynecologic malignancy other than endometrial cancer.
2. Current or untreated cervical, vaginal, or vulvar intraepithelial neoplasia or carcinoma.
3. History of total or subtotal hysterectomy, trachelectomy, radical trachelectomy, or pelvic radiotherapy.
4. Active lower genital tract bleeding.
5. Immunosuppressed state (e.g., HIV infection, status post organ transplantation).
6. Failure to undergo the planned hysteroscopic evaluation and follow-up within 1 year after the initial assessment.
7. Failed hysteroscopic procedure.
8. Any other condition that, in the opinion of the investigator, makes the participant unsuitable for inclusion in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This multicenter, prospective cohort study aims to enroll approximately 3,500 adult women in China who are at medium-to-high risk for endometrial cancer according to Chinese clinical consensus guidelines. The study population specifically includes two groups: 1) women who are scheduled for a diagnostic hysteroscopy due to these risk factors, and 2) women who are currently undergoing conservative treatment (such as progesterone therapy or endometrial ablation) for existing endometrial lesions and have not received chemotherapy. All participants must have an intact cervix and be willing to participate in follow-up assessments. Participants will be followed for up to 12 months, with the enrollment target set to observe at least 20 endpoint events (diagnosis of endometrial intraepithelial neoplasia or invasive cancer).
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of CISENDO Test | Baseline (at the time of initial hysteroscopy)
  The proportion of participants with histologically confirmed endometrial intraepithelial neoplasia (EIN) or invasive endometrial cancer who have a positive CISENDO test result at baseline.

SECONDARY OUTCOMES:
Dynamic Change in DNA Methylation Level | From baseline to 12 months
  The relative change in DNA methylation level (as measured by the CISENDO test) between baseline and follow-up visits (6 and 12 months) in participants undergoing surveillance.
Positive and Negative Predictive Values of CISENDO Test | Baseline
  The probability that participants with a positive test result truly have the disease (PPV), and the probability that those with a negative result truly do not have the disease (NPV), using histology as the gold standard.
Diagnostic Accuracy (Area Under the ROC Curve) | Baseline
  The overall diagnostic performance of the CISENDO test, evaluated by the Area Under the Receiver Operating Characteristic (ROC) Curve (AUC).
Comparison of Screening Strategies | Baseline
  Comparison of diagnostic performance metrics (sensitivity, specificity, PPV, NPV) between the CISENDO test and traditional diagnostic pathways (e.g., ultrasound findings leading to hysteroscopy).
Association of Methylation Level with Risk Stratification | Baseline
  The correlation between baseline DNA methylation levels and participants' clinical risk stratification according to Chinese consensus guidelines.

IPD SHARING:
Plan to Share IPD: Undecided